CLINICAL TRIAL: NCT05910970
Title: Adjuvant Tislelizumab With or Without Lenvatinib for Patients at High-risk of Hepatocellular Carcinoma Recurrence After Curative Resection or Ablation: a Multicentric, Prospective Study
Brief Title: Adjuvant Tislelizumab Plus Lenvatinib for Patients at High-risk of HCC Recurrence After Curative Resection or Ablation
Acronym: PREVENT-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENT-2
Record Dates: First submitted 2023-06-11; First posted 2023-06-20 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma; Recurrence; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant tislelizumab plus lenvatinib (Experimental): Patients at high-risk of hepatocellular carcinoma recurrence after curative resection or ablation will receive adjuvant tislelizumab plus lenvatinib treatment for six months, HCC recurrence, or unacceptable adverse events.
  Interventions: Drug: Adjuvant tislelizumab plus lenvatinib
- Adjuvant tislelizumab (Active Comparator): Patients at high-risk of hepatocellular carcinoma recurrence after curative resection or ablation will receive adjuvant tislelizumab treatment for six months, HCC recurrence, or unacceptable adverse events.
  Interventions: Drug: Adjuvant tislelizumab

INTERVENTIONS:
Drug: Adjuvant tislelizumab plus lenvatinib — Patients at high-risk of hepatocellular carcinoma recurrence after curative resection or ablation will receive adjuvant tislelizumab plus lenvatinib treatment for six months, HCC recurrence, or unacceptable adverse events.
  Arms: Adjuvant tislelizumab plus lenvatinib
Drug: Adjuvant tislelizumab — Patients at high-risk of hepatocellular carcinoma recurrence after curative resection or ablation will receive adjuvant tislelizumab treatment for six months, HCC recurrence, or unacceptable adverse events.
  Arms: Adjuvant tislelizumab

SUMMARY:
Though hepatic resection and ablation are the curative treatments for patients with hepatocellular carcinoma (HCC), the 5-years recurrence-free survival is lower than 30%. In recent years, several immune checkpoint inhibitors have been approved in advanced or unresectable HCC. No study about the safety and efficacy of adjuvant immune checkpoint inhibitors for patients with HCC after hepatectomy is reported.

DETAILED DESCRIPTION:
Hepatic resection and ablation are the best treatments for patients with early stage hepatocellular carcinoma (HCC) or selected intermediate or advanced disease. However, the postoperative 5-years recurrent rate is up to 70%, for whom recurrence is a major cause of death. In recent years, several immune checkpoint inhibitors have been approved in advanced HCC by official guidelines. At the same time, four randomizead controlled trials about adjvuant immune checkpoint inhibitors for postoperative HCC are ongoing. A prospective cohort study found adjuvant immune checkpoint inhibitors with or without tyrosine kinase inhibitors may improve recurrence-free survival of patients at high-risk of HCC recurrence after curative resection (DOI: 10.1200/JCO.2023.41.16_suppl.4119. Journal of Clinical Oncology 41, no. 16_suppl. 4119). Therefore, the investigators plan to compare the safety and efficacy of adjuvant Tislelizumab plus lenvatinib to Tislelizumab monotherapy for patients with high-risk factor of HCC recurrence after curative resection and ablation in a multicentric, prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years (inclusive);
* Diagnosis of HCC confirmed by postoperative histopathology;
* Underwent curative resection, as defined based on intra- and postoperative criteria;
* With high-risk factors of recurrence after curative treatment, based on preoperative radiological imaging or pathology reports indicating a tumor at least 5 cm in diameter, micro- or macrovascular invasion (Vp1/Vp2), satellite or multinodular tumors, and/or Grade 3/4 pathology;
* No residual cancer detected by radiological imaging in the liver within 8 weeks after curative resection;
* Child-Pugh 5-7 scores liver function;
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

* Received neoadjuvant immune checkpoint inhibitors or tyrosine kinase inhibitors before resection or ablation;
* A history of other malignancies;
* History of active autoimmune or immunodeficiency diseases;
* Concurrent cardiac, pulmonary, cerebral, or renal dysfunction;
* Loss to follow-up within six months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrene-free survival | 3 years
  Recurrene-free survival will be calculated using the Kaplan-Meier method, and differences between groups are assessed for significance using the log-rank test.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival will be calculated using the Kaplan-Meier method, and differences between groups are assessed for significance using the log-rank test.
Adverse events | 1 years
  Adverse events are expressed as number and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Hong Zhong, Ph.D, Principal Investigator — Guangxi Medical University Cancer Hospital
Locations (1):
- Jian-Hong Zhong, Nanning, China

IPD SHARING:
Plan to Share IPD: Yes
Data available on request due to privacy/ethical restrictions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study is completed and publication in a journal.

REFERENCES:
- [Background] Chen K, Wei W, Liu L, Deng ZJ, Li L, Liang XM, Guo PP, Qi LN, Zhang ZM, Gong WF, Huang S, Yuan WP, Ma L, Xiang BD, Li LQ, Zhong JH. Lenvatinib with or without immune checkpoint inhibitors for patients with unresectable hepatocellular carcinoma in real-world clinical practice. Cancer Immunol Immunother. 2022 May;71(5):1063-1074. doi: 10.1007/s00262-021-03060-w. Epub 2021 Sep 24. PMID 34559308
- [Background] Zhong JH, Ma L, Li LQ. Postoperative therapy options for hepatocellular carcinoma. Scand J Gastroenterol. 2014 Jun;49(6):649-61. doi: 10.3109/00365521.2014.905626. Epub 2014 Apr 10. PMID 24716523
- [Background] Hack SP, Spahn J, Chen M, Cheng AL, Kaseb A, Kudo M, Lee HC, Yopp A, Chow P, Qin S. IMbrave 050: a Phase III trial of atezolizumab plus bevacizumab in high-risk hepatocellular carcinoma after curative resection or ablation. Future Oncol. 2020 May;16(15):975-989. doi: 10.2217/fon-2020-0162. Epub 2020 Apr 30. PMID 32352320
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Background] Li L, Wu PS, Liang XM, Chen K, Zhang GL, Su QB, Huo RR, Xie RW, Huang S, Ma L, Zhong JH. Adjuvant immune checkpoint inhibitors associated with higher recurrence-free survival in postoperative hepatocellular carcinoma (PREVENT): a prospective, multicentric cohort study. J Gastroenterol. 2023 Oct;58(10):1043-1054. doi: 10.1007/s00535-023-02018-2. Epub 2023 Jul 14. PMID 37452107